CLINICAL TRIAL: NCT02374775
Title: Exploring the MEchanism of Plaque Rupture in Acute Coronary Syndrome Using Coronary CT Angiography and computationaL Fluid Dynamics (EMERALD)
Brief Title: Exploring the MEchanism of Plaque Rupture in Acute Coronary Syndrome Using Coronary CT Angiography and computationaL Fluid Dynamic
Acronym: EMERALD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: HeartFlow, Inc. (Industry); Kyoto University, Graduate School of Medicine (Other); Inje University (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other); Wakayama Medical University (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: NCT02374775
Record Dates: First submitted 2014-09-22; First posted 2015-03-02 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Plaque, Atherosclerotic; Rupture, Spontaneous
Keywords: axial plaque stress; pressure; pressure gradient; coronary plaque; plaque rupture; acute coronary syndrome; acute myocardial infarction; computational fluid dynamics; coronary computed tomography angiography; wall shear stress
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Plaque, Atherosclerotic; Rupture, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A (Culprit lesion): The plaque in the culprit vessel of acute myocardial infarction will be defined the Group A.
- Group B (Non-culprit lesion): The plaque in the non-culprit vessel of acute myocardial infarction will be defined as internal control, Group B.

SUMMARY:
The EMERALD trial is a multinational, multicenter study. The patients presented with AMI/definite evidence of plaque rupture and had underwent coronary CT angiography from 1 month to 2 year prior to the event will be retrospectively searched. Plaques in the non-culprit vessels will be regarded as internal control to the ruptured plaque in the culprit vessel.

DETAILED DESCRIPTION:
The mechanisms of plaque rupture have not been fully understood. Hemodynamic forces acting on the plaque, plaque vulnerability, and the interaction between two factors might be the most important mechanism to explain various feature and location of plaque rupture.

The objectives of the study are

1. To explore the interaction between hemodynamic forces measured by computational fluid dynamics (CFD) analysis and plaque vulnerability in culprit lesion of subsequent clinical events.
2. To build rupture risk scoring system, incorporating independent predictor for plaque rupture.

The EMERALD trial is a multinational and multicenter study. The patients presented with AMI/plaque rupture and had underwent coronary CT angiography from 1 month to 2 year prior to the event will be retrospectively searched. Plaques in the non-culprit vessels will be regarded as internal control to the ruptured plaque in the culprit vessel.

The enrollment criteria will be

1. Patients who presented with acute coronary syndrome with cardiac enzyme elevation (AMI)/plaque rupture.
2. Among those patients, the patients who underwent coronary CT angiography, regardless of the reason prior to the acute event will be searched. The time limit of coronary CT angiography will be 1 month ~ 2 year prior to the event.

The Computational Fluids Dynamics (CFD) and Fluid-Structural Interaction (FSI) simulation will be performed to comprehensively evaluate the total plaque forces and their interaction with the plaque.

The comparison groups will be defined as follows; The plaque in the culprit vessel of AMI will be defined the Group A. The plaque in the non-culprit vessel of AMI will be defined as internal control, Group B.

ELIGIBILITY:
Inclusion Criteria:

* Patients who experienced acute myocardial infarction from 2010-2014 whose diagnosis have confirmed by invasive coronary angiography with or without IVUS or OCT evaluation, and who underwent coronary CT angiography from 1 month to 2 year prior to the acute myocardial infarction event.

Exclusion Criteria:

* Acute coronary syndrome without cardiac enzyme elevation (unstable angina)
* Patients who did not underwent coronary CT angiography, 1 month to 2 years prior to the acute myocardial infarction
* Poor CT images (unable to reconstruct 3 dimensional coronary artery model)
* The time period between coronary CT angiography and acute myocardial infarction exceed more than 2 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who experienced acute myocardial infarction from 2010-2014 whose diagnosis have confirmed by invasive coronary angiography with or without IVUS or OCT evaluation, and who underwent coronary CT angiography from 1 month to 2 year prior to the acute myocardial infarction event. Acute coronary syndrome without cardiac enzyme elevation (unstable angina) will be excluded. The time limit of the coronary CT angiography prior to the event is from 1 month to 2 year. Participating center will perform abovementioned search process.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The difference of area under curve between prediction model with adverse plaque characteristics and model with adverse plaque characteristics and hemodynamic forces | from 1 month - 2 year
  Model 1 : percent diameter stenosis + adverse plaque characteristics defined by CT angiography Model 2 : percent diameter stenosis + adverse plaque characteristics defined by CT angiography + Hemodynamic forces defined by computational fluid dynamics
The difference of net reclassification index between prediction model with adverse plaque characteristics and model with adverse plaque characteristics and hemodynamic forces | from 1 month - 2 year
  Model 1 : percent diameter stenosis + adverse plaque characteristics defined by CT angiography Model 2 : percent diameter stenosis + adverse plaque characteristics defined by CT angiography + Hemodynamic forces defined by computational fluid dynamics

SECONDARY OUTCOMES:
The best cut-off value of axial plaque stress to induce plaque rupture. | from 1 month - 2 year
The threshold of the plaque vulnerability (Housefiled unit of the plaque on CT) to induce rupture. | from 1 month - 2 year
The independent predictors for the plaque rupture using generalized estimating equation, and the c-index of the predicting models. | from 1 month - 2 year
The validity of rupture risk score which constructed from the predicting model. | from 1 month - 2 year
The differences in other hemodynamic parameters for example, pressure gradient, delta pressure, FFRCT, average and peak wall shear stress between Group A and Group B. | from 1 month - 2 year
The association between axial plaque stress and the parameter reflecting plaque geometry (radius gradient). | from 1 month - 2 year
The differences in axial plaque stress between Group A and Group B | from 1 month - 2 year
The differences in plaque vulnerability (Housefiled unit of the plaque on CT) between Group A and Group B | from 1 month - 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Chair — Seoul National University Hospital; Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital; Joo Myung Lee, MD, MPH, Study Director — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Seoul national university hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After acceptance of first manuscript, the data will be shared upon request and permission of principal investigator and participants of the study

REFERENCES:
- [Derived] Lee JM, Choi G, Koo BK, Hwang D, Park J, Zhang J, Kim KJ, Tong Y, Kim HJ, Grady L, Doh JH, Nam CW, Shin ES, Cho YS, Choi SY, Chun EJ, Choi JH, Norgaard BL, Christiansen EH, Niemen K, Otake H, Penicka M, de Bruyne B, Kubo T, Akasaka T, Narula J, Douglas PS, Taylor CA, Kim HS. Identification of High-Risk Plaques Destined to Cause Acute Coronary Syndrome Using Coronary Computed Tomographic Angiography and Computational Fluid Dynamics. JACC Cardiovasc Imaging. 2019 Jun;12(6):1032-1043. doi: 10.1016/j.jcmg.2018.01.023. Epub 2018 Mar 14. PMID 29550316